CLINICAL TRIAL: NCT02484456
Title: An Investigation of the Antidepressant Effects of the Glycine Receptor Antagonist AV 101 (4-chlorokynurenine) in Major Depressive Disorder
Brief Title: Antidepressant Effects of the Glycine Receptor Antagonist AV-101 (4-chlorokynurenine) in Major Depressive Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 150151; 15-M-0151
Record Dates: First submitted 2015-06-26; First posted 2015-06-29 (Estimated); Results first posted 2022-03-02 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2019-12-03

CONDITIONS: Major Depression
Keywords: Major Depression; Glycine Receptor Antagonist; 4-chlorokynurenine; Treatment Resistant; Glutamatergic System
MeSH Terms: conditions — Depressive Disorder, Major | interventions — 4-chlorokynurenine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AV 101 (4-chlorokynurenine), then Placebo (Experimental): After a two-week drug-free period, participants received daily oral dose of AV 101 (4-chlorokynurenine) monotherapy 1,080mg/day for seven days, then dose increased to AV 101 1,440mg/day for next seven days followed by a two-week washout period; then crossover to placebo phase with daily dose of placebo pill for two weeks.
  Interventions: Drug: AV 101 (4-Chlorokynurenine); Other: Placebo Comparator
- Placebo, then AV 101 (4-chlorokynurenine) (Experimental): After a two-week drug-free period, participants received daily dose of placebo pill for two weeks followed by two-week washout period; then crossover to AV 101 treatment phase with daily oral dose of AV 101 (4-chlorokynurenine) monotherapy 1,080mg/day for seven days, then dose increased to AV 101 1,440mg/day for next seven days.
  Interventions: Drug: AV 101 (4-Chlorokynurenine); Other: Placebo Comparator

INTERVENTIONS:
Drug: AV 101 (4-Chlorokynurenine) — L-4-chlorokynurenine (4-Cl-KYN) was developed as a prodrug that is rapidly converted in vivo to its active metabolite 7-chlorokynurenic acid (7-Cl-KYNA), a well-characterized N-Methyl-D-aspartate receptor (NMDAR) antagonist at the glycine site.
  Other Names: 4-Cl-KYN
Other: Placebo Comparator — Placebo

SUMMARY:
Background:

- Drugs and talk therapy help treat depression, but these treatments usually take quite a bit of time to work. Ketamine is a fast-acting antidepressant, but it has side effects like unusual dreams and experiences. The drug AV-101 may have the same antidepressant effects but fewer side effects. Researchers want to see if it is effective and safe for people with major depressive disorder.

Objective:

- To see if the drug, AV-101 is safe and if it treats symptoms of major depressive disorder.

Eligibility:

- Adults ages 18-65 with major depression without psychotic features.

Design:

* Participants will be screened under a separate protocol.
* Participants will stay in the hospital for 12-14 weeks.
* Phase 1 (2-7 weeks): participants will stop taking their medicines then not take any for 2 weeks. They will have several scans and other procedures.
* Phase 2 (6-7 weeks): 2 weeks each of study drug and placebo once a day, with 2 weeks of no drugs in between.
* Participants will have:
* Physical exams
* Interviews
* Frequent blood collection. A needle will place a small plastic tube in the arm. Some blood samples will be taken through this tube.
* 2 spinal taps (optional). The back will be numbed. A needle will insert a catheter between back bones. That will be left in for up to 30 hours. Spinal fluid will be collected through it.
* 5 scans. Participants will lie in a machine with a magnetic field. The machine takes pictures of the brain and brain chemicals.
* At the end of the study, participants will have medical evaluation, questions, and blood tests. Some may continue treatment at the clinic.

DETAILED DESCRIPTION:
Objective

Modulation of the NMDA receptor (NMDAR) complex or other components of glutamatergic signaling is likely involved in improvement of depressive symptoms and related constructs/dimensions of observable behavior and neurobiological measures. Current standard monoaminergic pharmacological approaches for major depressive disorder (MDD) have proven to be only modestly effective during acute depressive episodes. We have systematically tested different glutamatergic modulators in patients with mood disorders in order to develop improved therapeutics. We found that the NMDAR antagonist ketamine produces rapid antidepressant effects in patients with treatment-resistant depression (in MDD and Bipolar Disorder). However, despite being highly efficacious, the proof of concept ketamine produces psychotomimetic effects.

In the present protocol, we aim to evaluate a new glutamate-mediated mechanism associated with antidepressant efficacy by targeting the glycine receptor within the NMDA receptor. Targeting the glycine co-agonist site of the (NMDA) receptor may bypass potential adverse effects that occur with ketamine without affecting the robust efficacy observed. This may then result in the glutamate surge that has been associated with the rapid acting antidepressant effects of ketamine.

The present Phase 2 proof-of-concept study is designed to evaluate the antidepressant effects of AV 101 (L-4-chlorokynurenine or 4-Cl- KYN) in MDD; this is a synthetic compound which is enzymatically converted into the selective glycine/NMDAR antagonist 7-chlorokynurenine (7-Cl-KYNA) after crossing the blood brain barrier (BBB) and then reaching brain glial cells. In animal models of depression, 4-Cl-KYNA (AV 101) induced acute and prolonged antidepressant-like effects without exhibiting ketamine-like side effects as determined by the drug discrimination, conditioned place preference, and pre-pulse inhibition tests.

We will also evaluate the neurobiological mechanisms involved in the antidepressant response to AV 101. We expect that this effect may modulate glutamate transmission and reverse the clinical symptoms of depression. The demonstration that a glycine-antagonist produces antidepressant effects without psychotomimetic side effects would support the therapeutic relevance of the glycine site of the NMDAR and could direct the development of novel drug targets for the treatment of depression.

Study Population

Twenty-five individuals with treatment-resistant major depressive disorder (MDD) will be included.

Design

Male and female patients, ages 18 to 65 years, with a diagnosis of MDD, currently in an episode of major depression, will be recruited for this study. This study will consist of a randomized, double-blind crossover administration of either the glycine receptor antagonist AV 101 (1,080 or 1,440 mg/day given orally) or placebo for 2 weeks. The study will assess the efficacy in improving overall depressive symptomatology and tolerability of AV 101 in treatment-resistant MDD. Other aims of the study include: 1) determining whether changes in brain neurochemicals (e.g. glutamate) and peripheral biomarkers obtained via MRS and cerebrospinal fluid (CSF) correlate with antidepressant response (decrease in Hamilton Depression Rating Scale (HDRS) total scores) to AV 101 in patients with treatment-resistant MDD, and 2) examine other potential biomarkers of response.

Outcome Measures

Primary: Hamilton Rating Scale (HDRS) total score.

Secondary: Proportion of subjects achieving remission (HDRS less than or greater than 7) and response (greater than or equal to 50% reduction from baseline in HDRS total score); change from baseline in Hamilton Anxiety Rating Scale (HAM-A), Montgomery-Asberg Depression Rating Scale (MADRS), and the Columbia Suicide Severity Rating Scale (C-SSRS) total scores. Surrogate biomarkers of drug effect/response include: changes in prefrontal glutamate levels measured with 7T H-MRS.

ELIGIBILITY:
* INCLUSION CRITERIA:
* 18 to 65 years of age.
* Subjects must have a level of understanding sufficient to agree to all required tests and examinations, sign an informed consent document and verify understanding. To verify this, subjects must score greater than or equal to 80% on the consent quiz.
* Subjects must fulfill Diagnostic and Statistical Manual (DSM)-IV or DSM-V criteria for MDD, single episode or recurrent without psychotic features, based on clinical assessment and confirmed by a structured diagnostic interview (SCID-P). Subjects must be experiencing a current major depressive episode of at least 4 weeks duration.
* Subjects must have an initial score of at least 18 on the HDRS at screening and at baseline of study phase I.
* Subjects must have a current or past history of lack of response to one adequate antidepressant trial (may be from the same chemical class) operationally defined using the modified-Antidepressant Treatment History Form (ATHF).

EXCLUSION CRITERIA:

* Current psychotic features or a diagnosis of schizophrenia or any other psychotic disorder as defined in the DSM-IV or DSM-V.
* Subjects with a history of DSM-IV drug or alcohol dependency or abuse (or alcohol use disorder per DSM-V),except for caffeine or nicotine dependence within the preceding 3 months.
* Head injury that results in loss of consciousness exceeding 5 minutes (for the imaging component of the study).
* Subjects with a DSM IV or DSM-V Axis II diagnosis of borderline or antisocial personality disorder.
* Pregnant or nursing women or women of child bearing potential not using at least 1 medically accepted means of contraception from the time of enrollment in the study until 1 month after completion of the second phase. Examples of medically accepted means of contraception include oral, injectable, or implant birth control, condom, diaphragm with spermicide, intrauterine devices (IUD), tubal ligation, abstinence or partner with vasectomy. .
* Serious, unstable illnesses including hepatic, renal, gastroenterologic, respiratory, cardiovascular (including ischemic heart disease), endocrinologic, neurologic, immunologic, or hematologic disease.
* Subjects with clinical hyperthyroidism or hypothyroidism.
* Subjects with one or more seizures without a clear and resolved etiology.
* Clinically significant abnormal laboratory tests.
* Treatment with a reversible monoamine oxidase inhibitor (MAOI) within 4 weeks of study phase II.
* Treatment with fluoxetine or aripiprazole within 5 weeks of study phase II.
* Treatment with any other disallowed concomitant medication or TMS 14 days before randomization.
* Treatment with clozapine or electroconvulsive therapy (ECT) within 1 month of randomization.
* Lifetime history of deep brain stimulation.
* Subjects who, in the Principal Investigator's judgment, pose a current serious suicidal or homicidal risk.
* Positive HIV test
* Contraindications to MRS (metal in body, claustrophobia, etc for imaging)
* No structured psychotherapy will be permitted during the total duration of the study. Subjects unable or unwilling to stop psychotherapy will be unable to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-10-14 (Actual); Primary Completion 2019-02-21 (Actual); Study Completion 2019-12-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos A Zarate, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Johnston JN, Yuan P, Kadriu B, Akula N, Quintanilla B, Peng S, Jones GH, Schulmann A, Yavi M, Henter ID, McMahon FJ, Kalynchuk LE, Zarate CA Jr, Caruncho HJ. Response of iPSC-derived neurons from individuals with treatment-resistant depression to (2 R,6 R)-hydroxynorketamine and reelin: an exploratory study. Transl Psychiatry. 2025 Nov 18;15(1):524. doi: 10.1038/s41398-025-03724-6. PMID 41257792
- [Derived] Park LT, Kadriu B, Gould TD, Zanos P, Greenstein D, Evans JW, Yuan P, Farmer CA, Oppenheimer M, George JM, Adeojo LW, Snodgrass HR, Smith MA, Henter ID, Machado-Vieira R, Mannes AJ, Zarate CA. A Randomized Trial of the N-Methyl-d-Aspartate Receptor Glycine Site Antagonist Prodrug 4-Chlorokynurenine in Treatment-Resistant Depression. Int J Neuropsychopharmacol. 2020 Jul 29;23(7):417-425. doi: 10.1093/ijnp/pyaa025. PMID 32236521
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2015-M-0151.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 22 participants signed consent. 3 participants withdrew before start of treatment leaving 19 participants starting.
Groups:
- Placebo, Then AV 101 (4-chlorokynurenine): After a two-week drug-free period, participants received daily dose of placebo pill for two weeks followed by two-week washout period; then crossover to AV 101 (4-chlorokynurenine) treatment phase with daily oral dose of AV 101 monotherapy 1,080mg/day for seven days, then dose increased to AV 101 1,440mg/day for next seven days.
Period: First Treatment Period: Week 1
Arm/Group | AV 101 (4-chlorokynurenine), Then Placebo | Placebo, Then AV 101 (4-chlorokynurenine)
Started | 10 | 9
Completed | 10 | 9
Not Completed | 0 | 0
Period: First Treatment Period: Week 2
Arm/Group | AV 101 (4-chlorokynurenine), Then Placebo | Placebo, Then AV 101 (4-chlorokynurenine)
Started | 10 | 9
Completed | 10 | 9
Not Completed | 0 | 0
Period: Washout Period
Arm/Group | AV 101 (4-chlorokynurenine), Then Placebo | Placebo, Then AV 101 (4-chlorokynurenine)
Started | 10 | 9
Completed | 10 | 8
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Second Treatment Period: Week 1
Arm/Group | AV 101 (4-chlorokynurenine), Then Placebo | Placebo, Then AV 101 (4-chlorokynurenine)
Started | 10 | 8
Completed | 9 | 7
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Period: Second Treatment Period: Week 2
Arm/Group | AV 101 (4-chlorokynurenine), Then Placebo | Placebo, Then AV 101 (4-chlorokynurenine)
Started | 9 | 7
Completed | 9 | 6
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AV 101 (4-chlorokynurenine), Then Placebo | Placebo, Then AV 101 (4-chlorokynurenine) | Total
Number analyzed (Participants) | 10 | 9 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 9 | 19
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 5 | 5 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 8 | 8 | 16
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 9 | 8 | 17
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Model Adjusted Means for Hamilton Depression Rating Score
Description: The Hamilton Depression Rating scale is a 17-item global measure of depressive symptoms on a 5-point scale ranging from 0 = not present to 4 = severe (full score values = 0,1,2,3,4). Some items rated on a scale of 0-2 (0, 1, 2) with 0 = not present to 2 = more severe. Total scores are a sum of the individual items. The maximum total score being 52 on the 17-point scale, and the minimum score being 0.Total scores of 0-7 are considered as being normal, 8-16 suggest mild depression, 17-23 moderate depression and scores over 24 are indicative of severe depression.
Time Frame: Post Dose Day 0
Population: The primary analysis compared active drug condition with placebo condition. Using within subject data (each person serving as their own control), we estimated means for drug, placebo and their difference at each time point. If outcome data were missing subsequent to a participant dropping out, their available data was included in the model.
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- AV 101 (4-chlorokynurenine): Participants received daily oral dose of AV 101 monotherapy 1,080mg/day for seven days, then 1,440mg/day for next seven days.
- Placebo: Participants received a daily oral dose of placebo pills for 2 weeks.
Arm/Group | AV 101 (4-chlorokynurenine) | Placebo
Number analyzed (Participants) | 19 | 19
score on a scale | 20.22 (0.68) | 20.56 (0.51)
Statistical Analysis 1: Comparison: AV 101 (4-chlorokynurenine) vs Placebo; Test type: Superiority; p = 0.68, Mixed Models Analysis; Mean Difference (Final Values) = 0.34, Standard Error of Mean 0.79

2. Primary Outcome: Model Adjusted Means for Hamilton Depression Rating Score
Description: as for outcome 1
Time Frame: Post Dose Day 1
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | AV 101 (4-chlorokynurenine) | Placebo
Number analyzed (Participants) | 19 | 19
score on a scale | 20.22 (0.58) | 20.06 (0.52)
Statistical Analysis 1: Comparison: AV 101 (4-chlorokynurenine) vs Placebo; Test type: Superiority; p = 0.83, Mixed Models Analysis; Mean Difference (Final Values) = -0.16, Standard Error of Mean 0.72

3. Primary Outcome: Model Adjusted Means for Hamilton Depression Rating Score
Description: as for outcome 1
Time Frame: Post Dose Day 2
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | AV 101 (4-chlorokynurenine) | Placebo
Number analyzed (Participants) | 19 | 19
score on a scale | 20.75 (0.62) | 20.41 (0.71)
Statistical Analysis 1: Comparison: AV 101 (4-chlorokynurenine) vs Placebo; Test type: Superiority; p = 0.71, Mixed Models Analysis; Mean Difference (Final Values) = -0.34, Standard Error of Mean 0.89

4. Primary Outcome: Model Adjusted Means for Hamilton Depression Rating Score
Description: as for outcome 1
Time Frame: Post Dose Day 3
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | AV 101 (4-chlorokynurenine) | Placebo
Number analyzed (Participants) | 19 | 19
score on a scale | 19.51 (0.72) | 20.74 (0.83)
Statistical Analysis 1: Comparison: AV 101 (4-chlorokynurenine) vs Placebo; Test type: Superiority; p = 0.25, Mixed Models Analysis; Mean Difference (Final Values) = 1.23, Standard Error of Mean 1.06

5. Primary Outcome: Model Adjusted Means for Hamilton Depression Rating Score
Description: as for outcome 1
Time Frame: Post Dose Day 7
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | AV 101 (4-chlorokynurenine) | Placebo
Number analyzed (Participants) | 19 | 19
score on a scale | 21.28 (0.70) | 20.43 (1.10)
Statistical Analysis 1: Comparison: AV 101 (4-chlorokynurenine) vs Placebo; Test type: Superiority; p = 0.51, Mixed Models Analysis; Mean Difference (Final Values) = -0.85, Standard Error of Mean 1.27

6. Primary Outcome: Model Adjusted Means for Hamilton Depression Rating Score
Description: as for outcome 1
Time Frame: Post Dose Day 13
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | AV 101 (4-chlorokynurenine) | Placebo
Number analyzed (Participants) | 19 | 19
score on a scale | 21.52 (1.13) | 19.69 (1.13)
Statistical Analysis 1: Comparison: AV 101 (4-chlorokynurenine) vs Placebo; Test type: Superiority; p = 0.26, Mixed Models Analysis; Mean Difference (Final Values) = -1.83, Standard Error of Mean 1.58

7. Secondary Outcome: Model Adjusted Means for Beck Depression Score
Description: The Beck Depression Inventory (BDI) is a 21-item measure of depression with each question on a 4-point scale ranging from 0=minimal to 3 = more severe (full list score values = 0,1,2,3). Total scores are a sum of individual items. The minimal depression = 0-13, mild depression = 14-19, moderate depression = 20-28, and severe depression = 29-63. The maximum score being 63 and the minimum possible score = 0.
Time Frame: Post Dose Day 0
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | AV 101 (4-chlorokynurenine) | Placebo
Number analyzed (Participants) | 19 | 19
score on a scale | 25.35 (0.79) | 25.79 (0.63)
Statistical Analysis 1: Comparison: AV 101 (4-chlorokynurenine) vs Placebo; Test type: Superiority; p = 0.67, Mixed Models Analysis; Mean Difference (Final Values) = 0.44, Standard Error of Mean 1.02

8. Secondary Outcome: Model Adjusted Means for Beck Depression Score
Description: as for outcome 7
Time Frame: Post Dose Day 1
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | AV 101 (4-chlorokynurenine) | Placebo
Number analyzed (Participants) | 19 | 19
score on a scale | 24.76 (0.84) | 24.75 (1.04)
Statistical Analysis 1: Comparison: AV 101 (4-chlorokynurenine) vs Placebo; Test type: Superiority; p = 0.99, Mixed Models Analysis; Mean Difference (Final Values) = -0.01, Standard Error of Mean 1.34

9. Secondary Outcome: Model Adjusted Means for Beck Depression Score
Description: as for outcome 7
Time Frame: Post Dose Day 2
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | AV 101 (4-chlorokynurenine) | Placebo
Number analyzed (Participants) | 19 | 19
score on a scale | 25.88 (0.67) | 26.14 (0.99)
Statistical Analysis 1: Comparison: AV 101 (4-chlorokynurenine) vs Placebo; Test type: Superiority; p = 0.83, Mixed Models Analysis; Mean Difference (Final Values) = 0.26, Standard Error of Mean 1.20

10. Secondary Outcome: Model Adjusted Means for Beck Depression Score
Description: as for outcome 7
Time Frame: Post Dose Day 3
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | AV 101 (4-chlorokynurenine) | Placebo
Number analyzed (Participants) | 19 | 19
score on a scale | 25.64 (0.69) | 24.64 (1.35)
Statistical Analysis 1: Comparison: AV 101 (4-chlorokynurenine) vs Placebo; Test type: Superiority; p = 0.51, Mixed Models Analysis; Mean Difference (Final Values) = -1.00, Standard Error of Mean 1.51

11. Secondary Outcome: Model Adjusted Means for Beck Depression Score
Description: as for outcome 7
Time Frame: Post Dose Day 7
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | AV 101 (4-chlorokynurenine) | Placebo
Number analyzed (Participants) | 19 | 19
score on a scale | 25.82 (1.13) | 24.22 (1.35)
Statistical Analysis 1: Comparison: AV 101 (4-chlorokynurenine) vs Placebo; Test type: Superiority; p = 0.37, Mixed Models Analysis; Mean Difference (Final Values) = -1.60, Standard Error of Mean 1.76

12. Secondary Outcome: Model Adjusted Means for Beck Depression Score
Description: as for outcome 7
Time Frame: Post Dose Day 13
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | AV 101 (4-chlorokynurenine) | Placebo
Number analyzed (Participants) | 19 | 19
score on a scale | 25.86 (1.09) | 23.84 (1.55)
Statistical Analysis 1: Comparison: AV 101 (4-chlorokynurenine) vs Placebo; Test type: Superiority; p = 0.29, Mixed Models Analysis; Mean Difference (Final Values) = -2.02, Standard Error of Mean 1.89

13. Secondary Outcome: Model Adjusted Means for Hamilton Anxiety Rating Score
Description: The Hamilton Anxiety Rating Scale (HAM-A) is a 14-item global measure of anxiety symptoms. Each item is scored on a scale of 0 (not present) to 4 (severe) (full score list = 0,1,2,3,4), with a total score range of 0-56 (0 = minimum score and 56 = maximum), where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe. Total scores are a sum of individual items.
Time Frame: Post Dose Day 0
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | AV 101 (4-chlorokynurenine) | Placebo
Number analyzed (Participants) | 19 | 19
score on a scale | 15.71 (0.56) | 16.20 (0.72)
Statistical Analysis 1: Comparison: AV 101 (4-chlorokynurenine) vs Placebo; Test type: Superiority; p = 0.60, Mixed Models Analysis; Mean Difference (Final Values) = 0.49, Standard Error of Mean 0.92

14. Secondary Outcome: Model Adjusted Means for Hamilton Anxiety Rating Score
Description: as for outcome 13
Time Frame: Post Dose Day 1
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | AV 101 (4-chlorokynurenine) | Placebo
Number analyzed (Participants) | 19 | 19
score on a scale | 17.30 (0.61) | 16.67 (0.75)
Statistical Analysis 1: Comparison: AV 101 (4-chlorokynurenine) vs Placebo; Test type: Superiority; p = 0.53, Mixed Models Analysis; Mean Difference (Final Values) = -0.63, Standard Error of Mean 0.98

15. Secondary Outcome: Model Adjusted Means for Hamilton Anxiety Rating Score
Description: as for outcome 13
Time Frame: Post Dose Day 2
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | AV 101 (4-chlorokynurenine) | Placebo
Number analyzed (Participants) | 19 | 19
score on a scale | 17.83 (0.55) | 17.66 (0.94)
Statistical Analysis 1: Comparison: AV 101 (4-chlorokynurenine) vs Placebo; Test type: Superiority; p = 0.88, Mixed Models Analysis; Mean Difference (Final Values) = -0.17, Standard Error of Mean 1.10

16. Secondary Outcome: Model Adjusted Means for Hamilton Anxiety Rating Score
Description: as for outcome 13
Time Frame: Post Dose Day 3
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | AV 101 (4-chlorokynurenine) | Placebo
Number analyzed (Participants) | 19 | 19
score on a scale | 16.48 (0.65) | 17.87 (0.62)
Statistical Analysis 1: Comparison: AV 101 (4-chlorokynurenine) vs Placebo; Test type: Superiority; p = 0.13, Mixed Models Analysis; Mean Difference (Final Values) = 1.40, Standard Error of Mean 0.91

17. Secondary Outcome: Model Adjusted Means for Hamilton Anxiety Rating Score
Description: as for outcome 13
Time Frame: Post Dose Day 7
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | AV 101 (4-chlorokynurenine) | Placebo
Number analyzed (Participants) | 19 | 19
score on a scale | 18.42 (0.74) | 17.25 (1.06)
Statistical Analysis 1: Comparison: AV 101 (4-chlorokynurenine) vs Placebo; Test type: Superiority; p = 0.38, Mixed Models Analysis; Mean Difference (Final Values) = -1.17, Standard Error of Mean 1.30

18. Secondary Outcome: Model Adjusted Means for Hamilton Anxiety Rating Score
Description: as for outcome 13
Time Frame: Post Dose Day 13
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | AV 101 (4-chlorokynurenine) | Placebo
Number analyzed (Participants) | 19 | 19
score on a scale | 18.33 (0.81) | 16.28 (0.97)
Statistical Analysis 1: Comparison: AV 101 (4-chlorokynurenine) vs Placebo; Test type: Superiority; p = 0.12, Mixed Models Analysis; Mean Difference (Final Values) = -2.05, Standard Error of Mean 1.26

19. Secondary Outcome: Model Adjusted Means for Montgomery-Asberg Depression Rating Score
Description: The Montgomery-Asberg Depression Rating Scale (MADRS) is a 10-item global measure evaluating core symptoms of depression. Questions concern how the patient has felt over the past week. Each item is rated on a scale from 0 to 6, with 0 being "normal/not present" and 6 being "extreme" (full score list = 0,1,2,3,4,5,6). Maximum score = 60, minimum score = 0. Total scores are a sum of the individual items.
Time Frame: Post Dose Day 0
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | AV 101 (4-chlorokynurenine) | Placebo
Number analyzed (Participants) | 19 | 19
score on a scale | 29.28 (0.62) | 29.48 (0.76)
Statistical Analysis 1: Comparison: AV 101 (4-chlorokynurenine) vs Placebo; Test type: Superiority; p = 0.84, Mixed Models Analysis; Mean Difference (Final Values) = 0.20, Standard Error of Mean 0.98

20. Secondary Outcome: Model Adjusted Means for Montgomery-Asberg Depression Rating Score
Description: as for outcome 19
Time Frame: Post Dose Day 1
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | AV 101 (4-chlorokynurenine) | Placebo
Number analyzed (Participants) | 19 | 19
score on a scale | 28.75 (0.63) | 28.79 (1.06)
Statistical Analysis 1: Comparison: AV 101 (4-chlorokynurenine) vs Placebo; Test type: Superiority; p = 0.97, Mixed Models Analysis; Mean Difference (Final Values) = 0.05, Standard Error of Mean 1.23

21. Secondary Outcome: Model Adjusted Means for Montgomery-Asberg Depression Rating Score
Description: as for outcome 19
Time Frame: Post Dose Day 2
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | AV 101 (4-chlorokynurenine) | Placebo
Number analyzed (Participants) | 19 | 19
score on a scale | 29.51 (0.48) | 29.84 (1.30)
Statistical Analysis 1: Comparison: AV 101 (4-chlorokynurenine) vs Placebo; Test type: Superiority; p = 0.81, Mixed Models Analysis; Mean Difference (Final Values) = 0.33, Standard Error of Mean 1.39

22. Secondary Outcome: Model Adjusted Means for Montgomery-Asberg Depression Rating Score
Description: as for outcome 19
Time Frame: Post Dose Day 3
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | AV 101 (4-chlorokynurenine) | Placebo
Number analyzed (Participants) | 19 | 19
score on a scale | 29.85 (0.71) | 30.81 (1.10)
Statistical Analysis 1: Comparison: AV 101 (4-chlorokynurenine) vs Placebo; Test type: Superiority; p = 0.47, Mixed Models Analysis; Mean Difference (Final Values) = 0.96, Standard Error of Mean 1.31

23. Secondary Outcome: Model Adjusted Means for Montgomery-Asberg Depression Rating Score
Description: as for outcome 19
Time Frame: Post Dose Day 7
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | AV 101 (4-chlorokynurenine) | Placebo
Number analyzed (Participants) | 19 | 19
score on a scale | 30.45 (0.89) | 28.64 (1.67)
Statistical Analysis 1: Comparison: AV 101 (4-chlorokynurenine) vs Placebo; Test type: Superiority; p = 0.35, Mixed Models Analysis; Mean Difference (Final Values) = -1.82, Standard Error of Mean 1.89

24. Secondary Outcome: Model Adjusted Means for Montgomery-Asberg Depression Rating Score
Description: as for outcome 19
Time Frame: Post Dose Day 13
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | AV 101 (4-chlorokynurenine) | Placebo
Number analyzed (Participants) | 19 | 19
score on a scale | 29.70 (1.05) | 27.06 (1.25)
Statistical Analysis 1: Comparison: AV 101 (4-chlorokynurenine) vs Placebo; Test type: Superiority; p = 0.12, Mixed Models Analysis; Mean Difference (Final Values) = -2.63, Standard Error of Mean 1.63

ADVERSE EVENTS:
Time Frame: 3 months
Groups:
- AV 101 (4-chlorokynurenine) 1,080 mg for 1 Week: Daily oral dose of AV 101 (4-chlorokynurenine) monotherapy 1,080mg/day for seven days
- AV 101 (4-chlorokynurenine) 1,440 mg for 1 Week: Daily oral dose of AV 101 (4-chlorokynurenine) monotherapy 1,440 mg/day for seven days
- Placebo 2 Weeks: Daily dose of placebo pill for two weeks
Arm/Group | AV 101 (4-chlorokynurenine) 1,080 mg for 1 Week | AV 101 (4-chlorokynurenine) 1,440 mg for 1 Week | Placebo 2 Weeks
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 1/19 | 1/19 | 0/19
Other Adverse Events (participants affected / at risk) | 9/19 | 7/19 | 6/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AV 101 (4-chlorokynurenine) 1,080 mg for 1 Week (N=19) | AV 101 (4-chlorokynurenine) 1,440 mg for 1 Week (N=19) | Placebo 2 Weeks (N=19)
Cerebrospinal fluid leakage (Injury, poisoning and procedural complications) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Speech disorder (Nervous system disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AV 101 (4-chlorokynurenine) 1,080 mg for 1 Week (N=19) | AV 101 (4-chlorokynurenine) 1,440 mg for 1 Week (N=19) | Placebo 2 Weeks (N=19)
Chest pain (Cardiac disorders) | 0 | 0 | 1
Eye irritation (Eye disorders) | 0 | 1 | 1
Vision blurred (Eye disorders) | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Cold sweat (General disorders) | 0 | 1 | 0
Decreased appetite (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 1
Irritability (General disorders) | 2 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 3
Advanced sleep phase (Nervous system disorders) | 1 | 0 | 2
Headache (Nervous system disorders) | 5 | 0 | 3
Insomnia (Nervous system disorders) | 3 | 0 | 2
Memory impairment (Nervous system disorders) | 2 | 1 | 1
Motor dysfunction (Nervous system disorders) | 1 | 0 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1
Sedation (Nervous system disorders) | 3 | 1 | 0
Sensory loss (Nervous system disorders) | 0 | 0 | 2
Sleep phase rhythm disturbance (Nervous system disorders) | 0 | 1 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pharyngitis (Gastrointestinal disorders) | 1 | 0 | 0
Reflux gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-15): https://cdn.clinicaltrials.gov/large-docs/56/NCT02484456/Prot_SAP_000.pdf